CLINICAL TRIAL: NCT04056052
Title: Mind the Gap! A Randomized Comparison Trial Examining the Impact of a Family-based Cooking Workshop on Vegetable Consumption, Self-efficacy and Willingness to Try of Children and Their Parents
Brief Title: A Randomized Comparison Trial Examining the Impact of a Family-based Cooking Workshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Sam Liu, Assistant Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UVic2012SCT
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Diet Habit
Keywords: Children; Family-based intervention
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Activity Only (Sham Comparator): Over the 8-week project, families were asked to try eight different vegetable recipes from a choice of 12. All family members could participate in the home activities as the families wished. Families were also asked to complete a weekly recipe cooking tracking sheet.
  Interventions: Behavioral: Mind the Gap: Home Activity Only
- Home Activity + cooking Workshop (Active Comparator): The 8-week cooking workshop condition incorporated all of the home activities previously described, however, this cohort also participated in two, two-hour cooking workshops held at a local cooking school.
  Interventions: Behavioral: Mind the Gap: Home Activity + cooking Workshop

INTERVENTIONS:
Behavioral: Mind the Gap: Home Activity Only — The primary focus of the home activity program was based on collaborative parent-child cooking activities which the families undertook themselves at home. There were two key tasks: the first was to add one extra vegetable to the evening meal each day, the second was to select, prepare and cook one recipe from the cook book each week.
  Arms: Home Activity Only
Behavioral: Mind the Gap: Home Activity + cooking Workshop — The main purpose of these workshops was to provide hands-on successful food preparation and cooking experiences for the families and several opportunities to taste new vegetable-based recipes as well as promoting knowledge of cost and healthy eating. Children and their parents were then encouraged to take whatever was learned and apply it at home.
  Arms: Home Activity + cooking Workshop

SUMMARY:
Increasing fruit and vegetable intake is important to health but children's vegetable intake remains low. In younger age groups parents act as gatekeepers by providing access, availability, persuasion and modelling. This study aimed to enhance parent vegetable serving behaviour and child vegetable intake through an 8-week social cognitive theory-based family cooking program.

ELIGIBILITY:
Inclusion Criteria:

* a family unit consisting of at least one parent and one child
* parents aged between 25 and 55 years of age
* children aged between nine and 13 years of age.

Exclusion Criteria:

* ability to comprehend English
* Participation of both the parent and the child

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Parent Food Serving Frequency | 7 days
  The scale included nine items assessing fruit and vegetable servings including potatoes and 100% fruit juice. Responses were on a 9 point likert scale ranging from 0 which represented never to 9 which represented serving vegetables more than 5 times/per day. For the entire scale, a conversion factor was used to transform responses into average daily servings for each item. To determine parental fruit and vegetable serving behavior, serving habits at breakfast, lunch and dinner for both fruits and vegetables were summed together to provide a score for overall number of servings served. This was also split into the specific number of fruits or vegetables served.
Child Food Frequency Questionnaire | 7 days
  A Food Frequency Questionnaire for children was used to measure typical weekly intake of fruit and vegetables including two items that addressed fried and white potato intake and one item that addressed 100% juice consumption. The scale was adapted from the US national cancer institute quick scan of fruit and vegetable and validated by Baranowski and colleagues [41]. The questionnaire consisted of nine items formatted as a 9 point likert scale whereby 0 represented never consumed and 9 represented consuming vegetables more than five times a day. A conversion factor was used to transform responses into average daily servings for each item, thus higher scores reflected the food choice being eaten more often on a daily basis. Similarly, assessing fruit and vegetable intake was determined by tallying the number of servings consumed across breakfast, lunch and dinner for both fruit and vegetables collectively and independently.

SECONDARY OUTCOMES:
Cooking confidence (Parent and Child) | 7 days
  Confidence in parents' general cooking/culinary abilities was also measured using part of a scale developed by Barton, Wrieden and Anderson [43] combined with two original items that were added to specifically address kitchen skills. Items addressing cooking confidence included questions such as, "how confident do you feel about measuring ingredients." The scale used a 7-point likert scale from "very unconfident" to "very confident". The six items were summed together to produce an overall score ranging from 6 to 42 with higher scores indicating greater sense of cooking self-efficacy. Scale reliability analysis showed that this measure also had good internal consistency (Cronbach's α = 0.95).
Outcome Expectations (Parent and Child) | 7 days
  13 items were used to assess outcome expectancies across three areas of known barriers; 1) expectations about taste, 2) expectations about the cost of healthy eating and 3) expectations about the level of effort required to prepare healthy meals. Each item represented a 7-point likert scale ranging from "strongly disagree" to "strongly agree." Items addressing barriers to healthy eating included statements such as, "it is quite expensive to follow a healthy diet." The overall scale was scored by summing all items and items that were negatively worded were reversed scored. Higher scores represented a lower perception of barriers to healthy eating. Scale reliability analysis revealed the overall scale to have good internal consistency (Cronbach's α = 0.79) while the subscales of taste, cost and effort had reliabilities of 0.72, 0.69, 0.68 respectively.
Exposure, Food Neophobia and Tast Preference (Parent and Child) | 7 days
  A previously validated and internally consistent (Cronbach's α = 0.88) version of a food neophobia scale for children [7,14,45] was used to measure parent fruit and vegetable neophobia with one modification. The item "when my parent asks me to eat…" on the children's scale was changed to "when my partner asks me to eat…" on the parent's scale. The food neophobia scale included eight items with all responses falling within a 7-point likert scale read from "strongly disagree" to "strongly agree". A total score was calculated by summing all eight items for a range of scores from 8 to 56. Higher scores represented a greater willingness to try new fruits and vegetables.

CONTACTS AND LOCATIONS:
Overall Officials: Patti-Jean Naylor, PhD, Principal Investigator — University of Victoria
Locations (1):
- University of Victoria, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided